CLINICAL TRIAL: NCT00275691
Title: Evaluation of Respiratory Specimens for Bacterial and Viral Pathogens by Real-Time PCR
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Franklin R Cockerill, MD, Mayo Clinic
Other Study IDs: 2354-02
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2010-01-18 (Estimated); Status verified 2010-01

CONDITIONS: Cough; Fever
MeSH Terms: conditions — Cough; Fever

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Community acquired pneumonia(CAP) is a common cause of morbidity and mortality. The diagnosis of CAP from the microbiology perspective has been challenging. Recent reports suggest the utility of real-time PCR for rapid and accurate diagnoses of these pathogens. Real-Time PCR tests, using the LightCycler instrument, will be performed on excess or additional specimens after extraction of nucleic acid.

DETAILED DESCRIPTION:
Excess patient specimens normally collected for routine microbiologic testing for CAP and in some cases additional specimens (i.e.,blood, urine, throat swab) will be evaluated using real-time PCR tests developed in our laboratory. Specimens will be performed on patients suspect for CAP. Test will be directed at variety of pathogens including but not limited to M.pneumoniae, C. pneumoniae, Legionella pneumophila, Streptococcus pneumoniae, B. pertussis, influenza viruses, adenovirus, and metapneumovirus. The ultimate goal is to have a panel of highly accurate and rapid (same day) tests that can be orderable and performed in short period time for CAP cases.

Real-Time PCR tests, using the LightCycler instrument, will be performed on excess or additional specimens after extraction of nucleic acid. Real-time PCR tests, using the LightCycler instrument, will be performed on excess or additional specimens after extraction nucleic acid. These tests will include the organisms listed above. As nucleic acid extracts will be archived, other pathogens can be tested in the future should we develop additional real-time PCR tests. All results obtained by real-time PCR will be compared to results for conventional testing as listed above. Sensitivity, specificity and predictive values will be calculated. In cases where discordant results occur, additional PCR testing and or medical history review will be conducted.

ELIGIBILITY:
Greater than 18 years of age. Cough present greater than one day and a history of fever and chills or documented fever in the Emergency Department

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Greater than 18 years of age. Cough present greater than one day and a history of fever and chills or documented fever in the Emergency Department
Sampling Method: Probability Sample
Enrollment: 867 (Actual)
Dates: Start 2005-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franklin R. Cockerill, III, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States